CLINICAL TRIAL: NCT03526835
Title: Phase 1/2 Dose Escalation and Cohort Expansion Study Evaluating MCLA-158 (Petosemtamab) as Single Agent or in Combination in Advanced Solid Tumors
Brief Title: A Study of Bispecific Antibody MCLA-158 in Patients With Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Merus B.V. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MCLA-158-CL01; 2017-004745-24 (EudraCT Number); 2024-513627-16-01 (EU CTIS Number)
Record Dates: First submitted 2018-04-04; First posted 2018-05-16 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2025-01

CONDITIONS: Advanced/Metastatic Solid Tumors; Colorectal Cancer; Gastric Cancer; Gastroesophageal-junction Cancer; NSCLC; HNSCC; Head and Neck Squamous Cell Carcinoma; Esophageal Cancer
Keywords: Bispecific antibody; First-in-human; MCLA-158; Antibodies; Bispecific; immunologic factors; Cytokines; EGFR; LGR5
MeSH Terms: conditions — Colorectal Neoplasms; Stomach Neoplasms; Squamous Cell Carcinoma of Head and Neck; Esophageal Neoplasms | interventions — pembrolizumab; Folfox protocol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- MCLA-158 (Experimental): In Part 1, the dose escalation phase, patients with metastatic CRC will receive escalating doses of MCLA-158 (every 2 weeks) until MTD or RP2D is reached. Each Cycle is 28 days. Single agent treatment.
  In Part 2, the expansion phase, participants with metastatic CRC and certain other solid tumors will receive intravenous infusion of MCLA-158 at the recommended Phase II dose (RP2D) every 2 weeks, at Day 1 and Day 15. The duration of each treatment cycle is 28 days. In addition, in the expansion phase, one randomized cohort will evaluate 2 doses (1100 mg and 1500 mg) of MCLA-158 in head and neck squamous cell carcinoma patients.
  Interventions: Drug: MCLA-158
- MCLA-158 + Pembrolizumab (Experimental): MCLA-158 in combination with pembrolizumab will be explored first in head and neck squamous cell carcinoma patients eligible to receive pembrolizumab as first-line monotherapy.
  Interventions: Combination Product: MCLA-158 + Pembrolizumab
- MCLA-158 + FOLFIRI combination chemotherapy (Experimental): MCLA-158 in combination with FOLFIRI will be explored in mCRC patients with up to 1 line of prior regimen.
  Interventions: Combination Product: MCLA-158 + FOLFIRI
- MCLA-158 + FOLFOX combination chemotherapy (Experimental): MCLA-158 in combination with FOLFOX will be explored in mCRC patients with up to 1 line of prior regimen.
  Interventions: Combination Product: MCLA-158 + FOLFOX

INTERVENTIONS:
Drug: MCLA-158 — full-length IgG1 bispecific antibody targeting EGFR and LGR5
  Other Names: petosemtamab
  Arms: MCLA-158
Combination Product: MCLA-158 + Pembrolizumab — MCLA-158 in combination with pembrolizumab will be explored first in HNSCC patients eligible to receive pembrolizumab as first-line monotherapy.
  Other Names: petosemtamab
  Arms: MCLA-158 + Pembrolizumab
Combination Product: MCLA-158 + FOLFIRI — MCLA-158 in combination with FOLFIRI will be explored in mCRC patients with up to 1 line of prior regimen.
  Other Names: petosemtamab
  Arms: MCLA-158 + FOLFIRI combination chemotherapy
Combination Product: MCLA-158 + FOLFOX — MCLA-158 in combination with FOLFOX will be explored in mCRC patients with up to 1 line of prior regimen.
  Other Names: petosemtamab
  Arms: MCLA-158 + FOLFOX combination chemotherapy

SUMMARY:
This is a Phase 1/2 open-label, multi-center, multi-national study with an initial dose escalation part to determine the recommended Phase II dose (RP2D) of MCLA-158 single agent in patients with mCRC.

The dose escalation part has been completed and the RP2D will be further evaluated in an expansion part of the study. Cohorts of selected solid tumor indications for which there is evidence of EGFR dependency and potential sensitivity to EGFR inhibition will be evaluated including head and neck cancer and metastatic colorectal cancer (mCRC).

The study will further assess the safety, tolerability, PK, PD, immunogenicity, and anti-tumor activity of MCLA-158 in monotherapy or in combination with other therapies.

DETAILED DESCRIPTION:
Study Design:

This open label, multicenter, first-in-human study consists of 2 parts. Part 1 is a dose escalation to find the recommended Phase II dose (RP2D) of MCLA-158 studying patients with metastatic colorectal cancer (mCRC). Enrollment in the dose escalation part has been completed.

In the dose expansion (single-agent cohorts) part of the study, the activity, safety, and tolerability of MCLA-158 at 1500 mg every 2 weeks (Q2W) (preliminary RP2D) as a single agent will be evaluated in cohorts of selected solid tumor indications with dependency on EGFR signaling. The most recently enrolled cohorts were in patients with head and neck squamous cell carcinoma (HNSCC). Enrollment into the HNSCC cohort of single-agent MCLA-158 for the treatment of patients with second/third line (2L/3L) HNSCC is closed. In the dose expansion part of the study, safety was also characterized at two dose levels in this setting. Other closed cohort indications included gastric/gastroesophageal junction adenocarcinoma (GEA) with EGFR amplification and/or high EGFR expression, esophageal carcinoma, and pancreatic adenocarcinoma. Enrollment is currently being explored in mCRC (RAS/RAF wild type) patients in the 3L/4L/5L setting.

Additionally, in the dose expansion (combination cohorts) part of the study, the activity, safety, and tolerability of MCLA-158 at 1500 mg Q2W will be evaluated in combination with other therapies. Enrollment in the combination cohort of treatment of MCLA-158 with pembrolizumab for the treatment of patients with first line (1L) HNSCC is closed. Additionally, two combination cohorts of MCLA-158 with FOLFIRI or with FOLFOX chemotherapy (i.e., 5-fluorouracil [5-FU], leucovorin, and irinotecan (FOLFIRI) or oxaliplatin (FOLFOX)) will be explored in mCRC (RAS/RAF wild type) patients in the 1L/2L setting. Other expansion cohorts may be considered for monotherapy or combination treatment in the future.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed solid tumors with evidence of metastatic or locally advanced disease not amenable to standard therapy with curative intent.
* A baseline fresh tumor sample (FFPE) from a metastatic or primary site (if safe/feasible).
* Amenable for biopsy (if safe/feasible).
* Measurable disease as defined by RECIST version 1.1 by radiologic methods.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Life expectancy ≥ 12 weeks, as per investigator.
* Left ventricular ejection fraction (LVEF) ≥ 50% by echocardiogram (ECHO) or multiple gated acquisition scan (MUGA).
* Adequate organ function
* Expansion cohorts: patients with locally advanced unresectable or metastatic disease for the following indications:

SINGLE AGENT:

* SECOND-/THIRD-LINE HNSCC PATIENTS (cohort closed to enrolment): patients who have progressed on or after, or are intolerant to, anti-PD-(L)1 therapy and platinum therapy as monotherapy or in combination with other agents and no previous exposure to EGFR inhibitors. Patients treated with platinum-containing therapy only in the adjuvant setting, or in the context of multimodal therapy for locally advanced disease should have disease progression within 6 months of the last dose of platinum containing therapy. Patients with no more than 2 prior lines of treatment in recurrent or metastatic disease.

  * Human papilloma virus (HPV) status determined by p16 immunohistochemistry (IHC) or molecular HPV test for all oropharyngeal tumors should be reported when available.
  * The eligible HNSCC primary tumor locations are oropharynx, oral cavity, hypopharynx, and larynx.
* 3L+ mCRC (cohort open to enrolment) patients must have:

  * No oncogenic missense mutations in KRAS, NRAS, BRAF, or EGFR ectodomain, and no HER2 (ERBB2) amplification, as detected in plasma by ctDNA NGS central testing performed during screening.
  * A microsatellite stable (MSS) tumor.

COMBINATION:

* FIRST-LINE HNSCC (cohort closed to enrolment): patients eligible to receive pembrolizumab as first-line monotherapy with tumors expressing programmed cell death protein ligand 1 (PD-L1), combined positive score (CPS) ≥1, as determined by a Food and Drug Administration (FDA) approved test in the US, or by an approved equivalent test in other countries; patients should not have previous systemic therapy administered in the recurrent or metastatic setting, although previous systemic therapy as part of multimodal treatment for locally advanced disease is allowed if ended ≥6 months prior to signing the ICF. The eligible HNSCC primary tumor locations are oropharynx, oral cavity, hypopharynx, and larynx. Previous treatments with anti PD-(L)1 or anti-EGFR therapies are not allowed.
* mCRC (cohorts open to enrolment): Patients should have been previously diagnosed with histologically or cytologically confirmed unresectable or metastatic adenocarcinoma of the colon or rectum. Patients must be RAS/RAF WT as determined using tumor tissue (primary or metastatic) by an appropriate tumor tissue based assay, to be confirmed by the sponsor, and must have an MSS tumor. Patients must be naive to prior anti-EGFR therapy.

  * Cohort to be treated with petosemtamab and FOLFIRI: patients may have received up to 1 prior chemotherapy regimen for the metastatic setting, consisting of 1L fluoropyrimidine-oxaliplatin-based chemotherapy ± bevacizumab.
  * Cohort to be treated with petosemtamab and FOLFOX: patients may have received up to 1 prior chemotherapy regimen in the metastatic setting consisting of 1L fluoropyrimidine-irinotecan-based chemotherapy ± bevacizumab.

Exclusion Criteria:

* Central nervous system metastases that are untreated or symptomatic, or require radiation, surgery, or continued steroid therapy to control symptoms within 14 days of study entry.
* Known leptomeningeal involvement.
* Participation in another clinical study or treatment with any investigational drug within 4 weeks prior to study entry.
* Any systemic anticancer therapy within 4 weeks or 5 half-lives whichever is shorter of the first dose of study treatment. For cytotoxic agents that have major delayed toxicity ( e.g. mitomycin C,nitrosoureas), or anticancer immunotherapies, a washout period of 6 weeks is required.
* Requirement for immunosuppressive medication (e.g. methotrexate, cyclophosphamide)
* Major surgery or radiotherapy within 3 weeks of the first dose of study treatment. Patients who received prior radiotherapy to ≥25% of bone marrow are not eligible, irrespective of when it was received.
* Persistent grade >1 clinically significant toxicities related to prior antineoplastic therapies (except for alopecia); stable sensory neuropathy ≤ grade 2 NCI-CTCAE v4.03 is allowed.
* History of hypersensitivity reaction to any of the excipients of petosemtamab, human proteins or any non-IMP treatment required for this study.
* Uncontrolled hypertension (systolic blood pressure [BP] > 150 mmHg and/or diastolic BP > 100 mmHg) with appropriate treatment or unstable angina.
* History of congestive heart failure of Class II-IV New York Heart Association (NYHA) criteria, or serious cardiac arrhythmia requiring treatment (except atrial fibrillation, paroxysmal supraventricular tachycardia).
* History of myocardial infarction within 6 months of study entry.
* History of prior malignancies with the exception of excised cervical intraepithelial neoplasia or nonmelanoma skin cancer, or curatively treated cancer deemed at low risk for recurrence with no evidence of disease for 3 years.
* Current dyspnea at rest of any origin, or other diseases requiring continuous oxygen therapy.
* Patients with a history of interstitial lung disease (e.g., pneumonitis or pulmonary fibrosis) or evidence of ILD on baseline chest computerized tomography (CT) scan.
* Current serious illness or medical conditions including, but not limited to uncontrolled active infection,clinically significant pulmonary, metabolic or psychiatric disorders.
* Patients with known infectious diseases:

  * Active hepatitis B infection ((hepatitis B surface antigen [HBsAg] positive) without receiving antiviral treatment.
  * Positive test for hepatitis C ribonucleic acid (HCV) RNA).
* Pregnant or breastfeeding patients; patients of childbearing potential must use highly effective contraception methods prior to study entry, for the duration of study participation, and for 6 months after the last dose of MCLA-158.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 523 (Estimated)
Dates: Start 2018-05-02 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Escalation: Number of patients with Dose Limiting Toxicities (DLTs) during Cycle 1 | 4 weeks
  Evaluation of the number and severity of participants with treatment related toxicities observed during the dose escalation.
Expansion (Single agent - randomized expansion in 2/3L Head and Neck cancer, and combination cohorts): Safety and tolerability: AEs and SAEs | 6-12 months
  Incidence, severity, and relationship of AEs and SAEs
Expansion (Single agent - randomized expansion in 2/3L Head and Neck cancer): Treatment discontinuations and dose modifications due to AEs | 6-12 months
  Treatment discontinuations due to AEs and dose modifications due to AEs
Expansion (single agent - randomized expansion in 2/3L Head and Neck cancer): Best overall response (BOR) | 36 months
  Evaluation of clinical benefit assessed by RECIST v1.1 determining Best overall response (BOR)
Expansion (Single agent - non-randomized, and combination cohorts): Objective response rate (ORR) | 36 months
  Evaluation of clinical benefit assessed by RECIST v1.1 determining objective response rate (ORR)
Expansion (single agent - randomized expansion in 2/3L Head and Neck cancer): exposure-safety relationship of petosemtamab administered at 1100 mg and 1500 mg: TEAEs | 8 weeks
  Incidence of TEAEs at Week 8

SECONDARY OUTCOMES:
Escalation & Expansion: Duration of response (DOR) | 36 months
  Evaluation of clinical benefit assessed by RECIST v1.1 determining duration of response (DOR)
Expansion: Progression Free Survival (PFS) | 36 months
  Evaluation of clinical benefit assessed by RECIST v1.1 determining progression free survival (PFS)
Expansion (mCRC combination cohorts): Progression Free Survival (PFS) rate at 4 months | 4 months
  Evaluation of clinical benefit assessed by RECIST v1.1 determining progression free survival (PFS) rate at 4 months
Expansion (Single agent - non-randomized cohorts): Overall survival (OS) | 36 months
  Evaluation of clinical benefit determining overall survival (OS)
Escalation & Expansion (single agent - non-randomized cohorts): Safety and tolerability: AEs and SAEs | up to 30 days post-last dose
  Incidence, severity, and relationship of AEs and SAEs
Escalation & Expansion (Single agent - non-randomized and Combination cohorts): Treatment discontinuations and dose modifications due to AEs | up to 30 days post-last dose
  Treatment discontinuations due to AEs and dose modifications due to AEs
Expansion (Single agent - randomized expansion in 2/3L Head and Neck cancer): exposure-efficacy relationship of petosemtamab administered at 1100 mg and 1500 mg: Target Lesions | 8 weeks
  Percentage change from baseline in sum of the diameters of target lesions at Week 8
Expansion (Single agent - randomized expansion in 2/3L Head and Neck cancer): exposure-safety relationship of petosemtamab administered at 1100 mg and 1500 mg: Grade 3-4 TEAEs | 8 weeks
  Incidence of Grade 3-4 TEAEs at Week 8
Expansion (Single agent - randomized expansion in 2/3L Head and Neck cancer): exposure-safety relationship of petosemtamab administered at 1100 mg and 1500 mg: IRR TEAEs | 8 weeks
  Incidence of IRR TEAEs at Week 8
Expansion (Single agent - randomized expansion in 2/3L Head and Neck cancer): exposure-safety relationship of petosemtamab administered at 1100 mg and 1500 mg : non-IRR TEAEs | 8 weeks
  Incidence of non-IRR TEAEs at Week 8
Escalation and Expansion: Safety and tolerability: laboratory values | 6-12 months
  Number of participants with abnormal laboratory tests results
Escalation and Expansion: Safety and tolerability: (ECG) | 6-12 months
  Number of participants with abnormal ECG readings
Escalation and Expansion: Safety and tolerability: vital signs | 6-12 months
  Number of participants with abnormal vital signs
Expansion (Single agent - randomized expansion in 2/3L Head and Neck cancer): Objective response rate (ORR) | 36 months
  Evaluation of clinical benefit assessed by RECIST v1.1 determining objective response rate (ORR)
Escalation & Expansion: Incidence of anti-drug antibodies against MCLA-158 | 36 months
  Number of participants with anti-drug antibodies against MCLA-158
Escalation: Cytokine Panel Expression Profile | 36 months
  Evaluation of the cytokine expression profile
Escalation & Expansion: End of infusion (EOI) plasma concentration [Ceoi] | 36 months
  End of infusion (EOI) plasma concentration [Ceoi] as measured from all individual plasma concentrations
Escalation & Expansion: Maximum plasma concentration [Cmax] | 36 months
  Maximum plasma concentration as measured from all individual plasma concentrations
Escalation & Expansion: Plasma concentration at 0 hours [C0h] | 36 months
  Plasma concentration at 0 hours [C0h] as measured from all individual plasma concentrations
Escalation & Expansion: Area under the concentration versus time curve from time zero to time t [AUC0-t] | 36 months
  Area under the concentration versus time curve from time zero to time t [AUC0-t]
Escalation & Expansion: Area under the concentration versus time curve [AUC0-∞] | 36 months
  Area under the concentration versus time curve [AUC0-∞]
Escalation & Expansion: Clearance of plasma [CL] | 36 months
  Clearance of plasma [CL]
Escalation & Expansion: Volume of distribution at steady state [Vss] | 36 months
  Volume of distribution at steady state [Vss]
Escalation & Expansion: Half-life [t1/2] | 36 months
  Half-life [t1/2]

CONTACTS AND LOCATIONS:
Overall Officials: Gianluca Laus, MD, Study Director — Merus B.V.
Locations (45):
- United States (23):
  - UCSD, La Jolla, California
  - USC Norris Comprehensive Cancer Center, Los Angeles, California
  - Sharp Healthcare, San Diego, California
  - Rocky Mountain Cancer Centers, Lone Tree, Colorado
  - Florida Cancer Specialists, Fort Myers, Florida
  - Sarah Cannon Research Institute (Lake Nona), Orlando, Florida
  - Massachusetts General Hospital - Dana Farber, Boston, Massachusetts
  - SSM Health Saint Louis University Hospital, St Louis, Missouri
  - Washington University School of Medicine at St Louis, St Louis, Missouri
  - Cayuga Medical Center, Ithaca, New York
  - Hematology-Oncology Associates of Central New York, Syracuse, New York
  - Cleveland Clinic, Cleveland, Ohio
  - Taylor Cancer Research Center, Maumee, Ohio
  - SSM OKC Hightower Clinical, Oklahoma City, Oklahoma
  - The University Of Tennessee Health Science Center, Memphis, Tennessee
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - Texas Oncology, Dallas, Texas
  - Oncology Consultants, Houston, Texas
  - Texas Oncology, Tyler, Texas
  - Utah Cancer Specialists, Salt Lake City, Utah
  - University of Utah Health Huntsman Cancer Hospital, Salt Lake City, Utah
  - Oncology & Hematology Associates of Southwest Virginia, Roanoke, Virginia
  - Cancer Care Northwest, Spokane, Washington
- Belgium (4):
  - Cliniques universitaires Saint-Luc, Brussels
  - Institut Jules Bordet, Brussels
  - UZ Gent, Ghent
  - Chu Ucl Namur Site De Sainte-Elisabeth, Namur
- France (8):
  - Hopital Saint Andre, CHU Bordeaux, Bordeaux
  - Centre Leon Berard, Lyon
  - Hopital La Timone, Marseille
  - Institut Régional du Cancer de Montpellier, Montpellier
  - Centre Antoine Lacassagne, Nice
  - Institut Curie, Paris
  - Institut Gustave Roussy, Paris
  - Centre Henri Becquerel, Rouen
- Netherlands (3):
  - NKI - Antoni van Leeuwenhoek, Amsterdam
  - UMC Radboud, Nijmegen
  - UMC Utrecht, Utrecht
- Spain (5):
  - Vall d'Hebron, Barcelona
  - Hospital 12 de Octubre, Madrid
  - Clinica Universidad de Navarra, Pamplona
  - Hospital Universitario de Navarra, Pamplona
  - Instituto Valenciano de Oncologia, Valencia
- United Kingdom (2):
  - Cambridge University Hospitals NHS Foundation Trust, Cambridge
  - Sarah Cannon Research Institute, London

IPD SHARING:
Plan to Share IPD: No